CLINICAL TRIAL: NCT01755936
Title: The Role of Myocardial Fibrosis in Patients With Aortic Stenosis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/R/CAR/05
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2016-07

CONDITIONS: Aortic Stenosis
Keywords: Aortic Stenosis; Cardiac magnetic resonance imaging; Late Gadolinium enhancement; T1 mapping techniques; Replacement fibrosis; Diffuse interstitial fibrosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full blood count and renal panel will be measured.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls: Patients will undergo cardiac magnetic resonance imaging, echocardiography and 72 hour holter monitoring
  Interventions: Other: Cardiac Magnetic Resonance Imaging; Other: Echocardiography; Other: 72 hour Holter Monitor
- Aortic Stenosis patients: All patients who agreed to study will undergo cardiac magnetic resonance imaging, echocardiography and 72 hour holter monitoring
  Interventions: Other: Cardiac Magnetic Resonance Imaging; Other: Echocardiography; Other: 72 hour Holter Monitor

INTERVENTIONS:
Other: Cardiac Magnetic Resonance Imaging — For the evaluation of left ventricular volumes, function and mass. Also for the assessment of myocardial fibrosis based on the presence of delayed enhancement. Novel application of T1 mapping techniques will be evaluated.
Other: Echocardiography — Assessment of aortic stenosis severity. Also evaluate diastolic and systolic function.
Other: 72 hour Holter Monitor — This will enable us to detect abnormal heart rhythms which may be associated with myocardial fibrosis

SUMMARY:
Aortic stenosis is the most common adult valvular heart disease in the western world. Heart failure and sudden cardiac death are complications associated with aortic stenosis. In symptomatic individuals, valve replacement is often the only effective treatment. However, there are no good markers to identify patients who may benefit from early surgery before symptoms developed. The purpose of the study is to test the hypothesis that the presence heart muscle scarring on the cardiac magnetic resonance imaging may predict a worse outcome in patients with aortic stenosis, and thus may be helpful in identifying patients for early valve replacement.

DETAILED DESCRIPTION:
Congestive heart failure and sudden cardiac death are associated complications of aortic stenosis. Currently, the indications for valvular replacement are based on the valvular severity evaluated by echocardiography and the presence of symptoms. There is some evidence to suggest the presence of myocardial fibrosis is associated with a poor outcome in patients with aortic stenosis. The aim of this prospective study is to investigate the prognostic implications of myocardial fibrosis in patients with aortic stenosis. The presence of myocardial fibrosis will be identified by delayed enhancement with the cardiac magnetic resonance imaging at 3T. We will also be evaluating the application of T1 mapping techniques to detect diffuse myocardial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aortic stenosis
* Willing to undergo all investigations

Exclusion Criteria:

* Coexisting mitral valvular heart disease and aortic regurgitation (more than moderate severity)
* Active medical conditions: ongoing heart failure, infection
* Significant comorbidities: advanced malignancy with limited life expectancy
* Unable to give informed consent
* Contraindication for cardiac magnetic resonance imaging: impaired renal function, pacemaker, claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 240 individuals will be recruited. This includes 48 individuals who do not have aortic stenosis. A total of 192 individuals with aortic stenosis will be recruited:
  1. Mild aortic stenosis, n=48
  2. Moderate aortic stenosis, n=48
  3. Severe aortic stenosis, n=48
  4. Symptomatic aortic stenosis with planned valve replacement, n=48
Sampling Method: Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | 1 year
  Cardiovascular events defined as cardiovascular deaths, development of heart failure symptoms, and the need for aortic valve replacement.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD PhD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Derived] Vassiliou VS, Pavlou M, Malley T, Halliday BP, Tsampasian V, Raphael CE, Tse G, Vieira MS, Auger D, Everett R, Chin C, Alpendurada F, Pepper J, Pennell DJ, Newby DE, Jabbour A, Dweck MR, Prasad SK. A novel cardiovascular magnetic resonance risk score for predicting mortality following surgical aortic valve replacement. Sci Rep. 2021 Oct 12;11(1):20183. doi: 10.1038/s41598-021-99788-7. PMID 34642428
- [Derived] Everett RJ, Tastet L, Clavel MA, Chin CWL, Capoulade R, Vassiliou VS, Kwiecinski J, Gomez M, van Beek EJR, White AC, Prasad SK, Larose E, Tuck C, Semple S, Newby DE, Pibarot P, Dweck MR. Progression of Hypertrophy and Myocardial Fibrosis in Aortic Stenosis: A Multicenter Cardiac Magnetic Resonance Study. Circ Cardiovasc Imaging. 2018 Jun;11(6):e007451. doi: 10.1161/CIRCIMAGING.117.007451. PMID 29914867
- [Derived] Anand A, Chin C, Shah ASV, Kwiecinski J, Vesey A, Cowell J, Weber E, Kaier T, Newby DE, Dweck M, Marber MS, Mills NL. Cardiac myosin-binding protein C is a novel marker of myocardial injury and fibrosis in aortic stenosis. Heart. 2018 Jul;104(13):1101-1108. doi: 10.1136/heartjnl-2017-312257. Epub 2017 Dec 1. PMID 29196542
- [Derived] Kwiecinski J, Chin CWL, Everett RJ, White AC, Semple S, Yeung E, Jenkins WJ, Shah ASV, Koo M, Mirsadraee S, Lang CC, Mills N, Prasad SK, Jansen MA, Japp AG, Newby DE, Dweck MR. Adverse prognosis associated with asymmetric myocardial thickening in aortic stenosis. Eur Heart J Cardiovasc Imaging. 2018 Mar 1;19(3):347-356. doi: 10.1093/ehjci/jex052. PMID 28379401
- [Derived] Chin CWL, Everett RJ, Kwiecinski J, Vesey AT, Yeung E, Esson G, Jenkins W, Koo M, Mirsadraee S, White AC, Japp AG, Prasad SK, Semple S, Newby DE, Dweck MR. Myocardial Fibrosis and Cardiac Decompensation in Aortic Stenosis. JACC Cardiovasc Imaging. 2017 Nov;10(11):1320-1333. doi: 10.1016/j.jcmg.2016.10.007. Epub 2016 Dec 21. PMID 28017384